CLINICAL TRIAL: NCT04882696
Title: Evaluation of the Impact of Non-slip Socks on Motor Recovery in the Elderly An Open Label, Single-center, Randomized, Controlled Pilot Study
Brief Title: Evaluation of the Impact of Non-slip Socks on Motor Recovery in the Elderly
Acronym: CHARM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow recruitment
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHD 20-0059
Record Dates: First submitted 2021-04-29; First posted 2021-05-12 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Aging; Acute Care Unit; Fall Injury
Keywords: non slip socks; aging; rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- usual care with bare feet (No Intervention): patients will be treated barefoot during their stay
- specific care with anti-slip socks (Experimental): Patients in this group will wear non-slip socks
  Interventions: Other: Non-slip socks

INTERVENTIONS:
Other: Non-slip socks — Patients will wear non-slip socks during their hospitalization
  Arms: specific care with anti-slip socks

SUMMARY:
Some authors suggest a possible clinical interest of anti-slip socks. The scientific literature presents studies with methodological limitations. It is therefore not currently possible to judge the specific interest of anti-slip socks in an elderly hospitalized population.

The investigatorswould therefore like to know the interest of wearing non-slip socks in the management of these patients, and more particularly on the main objective of rehabilitation in geriatric physiotherapy: motor function.

DETAILED DESCRIPTION:
Some authors suggest a possible clinical interest of anti-slip socks. The scientific literature presents studies with methodological limitations, but above all a different population than the one the investigators are interested in. It is therefore not currently possible to judge the specific interest of anti-slip socks in an elderly hospitalized population.

Evaluating the value of these socks could allow to recommend them with solid data. Preventing this iatrogenic loss of autonomy would have a positive impact on the motor capacities of patients, a quicker and easier return home, and a reduction in health costs.

The investigators would therefore like to know the interest of wearing non-slip socks in the management of these patients, and more particularly on the main objective of rehabilitation in geriatric physiotherapy: motor function.

ELIGIBILITY:
Inclusion Criteria:

* Patient in Geriatric acute care or Post-Emergency Medicine,
* Patient 75 years and older,
* Patient requiring physiotherapy,
* Patient with a minimum of 7 days of physical therapy
* Patient arrived with unsuitable footwear (assessment at the discretion of the clinician: no back support, unsuitable size, etc.) or without footwear,
* Patient able to walk at least 10 m with or without technical assistance,
* Patient who has given oral consent
* Patient with social security coverage.

Exclusion Criteria:

* Inability to understand or perform study-specific clinical tests
* Known cognitive impairment, disease or condition that compromises comprehension of information or informed consent by the patient
* Blind patient
* Patient under guardianship or curatorship
* Patient participating in an interventional clinical research protocol that may alter the assessments of this protocol.
* Patient previously included in the Charm study
* Patient with an identified risk of being unable to wear socks or to walk barefoot within the next 7 days (need for compression stockings or socks, wound, excessive edema, orthostatic hypotension, other)

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-03-04 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Change from Baseline walking speed (start of physiotherapy treatment) at D8. | Day 8
  Change from Baseline walking speed at the patient's preferred speed over 10m between (start of physiotherapy treatment) at D8.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas RULLEAU, Principal Investigator — Departmental Hospital Center of Vendee
Locations (1):
- Centre Hospitalier Departemental Vende, La Roche-sur-Yon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rulleau T, Planche L, Dorion A, Soldani G, Blain C, Chapeleau C, Bleher Y, Da Silva C, Launeau N, Joguet E, Fevrier R, Decours R. Evaluation of the impact of non-slip socks on the motor recovery of elderly people in acute care hospitals: Protocol for a randomized, controlled trial study. PLoS One. 2023 May 1;18(5):e0283226. doi: 10.1371/journal.pone.0283226. eCollection 2023. PMID 37126507

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-28): https://cdn.clinicaltrials.gov/large-docs/96/NCT04882696/Prot_SAP_000.pdf